CLINICAL TRIAL: NCT00422760
Title: A 75 Year Old With Dyspnea a Case Report.Observational Study
Status: Completed | Type: Observational
Sponsor: Stanley Medical College (Other Government)
Other Study IDs: Boerhaave
Record Dates: First submitted 2007-01-13; First posted 2007-01-17 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2007-01

CONDITIONS: Esophageal Perforation
Keywords: esophageal perforation; COPD
MeSH Terms: conditions — Esophageal Perforation; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
Clinical Case report Of spontaneous esophageal perforation in a 75 year old man. He prsented with breathlessness and on investigation found to have esophageal perforation

DETAILED DESCRIPTION:
Boerhaave's syndrome represents a diagnostic dilemma for the physician. Boerhaave's syndrome is an uncommon condition where there is oesophageal rupture following forceful vomiting. We report a case of spontaneous rupture of the esophagus in 75-year-old male with chronic obstructive pulmonary disease who was referred to our hospital with acute onset of breathlessness. The absence of vomiting prior to presentation is the distinguishing feature of this particular case.

ELIGIBILITY:
Inclusion Criteria:

* male with esophageal perforation man with COPD

Exclusion Criteria:

* Iatrogenic perforation

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1
Dates: Start 2007-01; Study Completion 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: Tiroporur G Balachandar, McH, Principal Investigator — Stanley medicl college